CLINICAL TRIAL: NCT00349791
Title: A Study to Evaluate the Efficacy/Safety of Transdermal Testosterone for 24 Weeks in Naturally Menopausal Women With Hypoactive Sexual Desire Disorder on Oral Hormone Replacement Therapy.
Brief Title: Study to Assess the Efficacy/Safety of Transdermal Testosterone Patches in Naturally Menopausal Women With Low Libido
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Warner Chilcott (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2002006
Record Dates: First submitted 2006-07-07; First posted 2006-07-10 (Estimated); Last update posted 2013-04-17 (Estimated); Status verified 2013-04

CONDITIONS: Hypoactive Sexual Desire Disorder (HSDD)
Keywords: Natural Menopause
MeSH Terms: conditions — Sexual Dysfunctions, Psychological

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Placebo Comparator): placebo patch replaced twice a week for two years
  Interventions: Drug: Placebo patch
- 2 (Experimental): testosterone patch replaced twice a week for two years
  Interventions: Drug: Testosterone Transdermal System

INTERVENTIONS:
Drug: Testosterone Transdermal System — testosterone (300 mcg/day) patch replaced twice a week for two years
  Arms: 2
Drug: Placebo patch — placebo patch replaced twice a week for two years
  Arms: 1

SUMMARY:
This study is designed to evaluate efficacy and safety of a testosterone patch as treatment for low libido in naturally menopausal women who are taking estrogen or estrogen/progestin therapy.

DETAILED DESCRIPTION:
Naturally menopausal women with hypoactive sexual desire disorder (HSDD) were randomized into a 24-week, multicenter, multinational, double-blind (DB), parallel-group, placebo-controlled study. Patients were randomized to receive a placebo or testosterone transdermal system throughout the study. Safety was assessed by adverse events, lipids, serum chemistry with hepatic, renal and carbohydrate metabolism evaluation, and hematology. Physical exam including clinical assessments of facial hair and acne were monitored.

ELIGIBILITY:
Inclusion Criteria:

Eligible women must:

1. Be 40-70 years old and in generally good health
2. Be post-menopausal with no spontaneous periods for 1 year
3. Be receiving a stable dose of hormone replacement therapy for at least 3 months pror to screening with the intention of maintaining that regimen.
4. Be, in her own judgment, in a stable, monogamous sexual relationship that is perceived to be secure and communicative, for at least one year prior to study entry
5. Meet the criteria for having hypoactive sexual desire disorder

Exclusion Criteria:

Eligible women must not:

1. Have received androgen therapy at any time during the past 3 months (during the past 7 months if therapy was an investigational implantable product)
2. Be experiencing any chronic or acute life stress relating to any major life change
3. Be experiencing depression and/or receiving medication for such illness or disorder
4. Have current severe skin problems (such as severe or cystic acne) or allergy to adhesives (like the ones in bandages)
5. Have had a major illness, active gall bladder disease, or gynecological or breast surgery within the last 6 months
6. Have a history of breast, endometrial, or other gynecological cancer at any time before study participation or other cancer within the last 5 years
7. Have diabetes, a history of cerebrovascular disease, thrombo-embolic disorders, heart attack, or angina at any time before study participation or thrombophlebitis within the last 5 years
8. Have abnormal laboratory test results upon initial screening for this study
9. Have previously participated in a clinical trial within 30 days or received an investigational medication within 30 days

Ages: 40 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 549 (Actual)
Dates: Start 2002-06; Primary Completion 2003-10 (Actual); Study Completion 2003-10 (Actual)

PRIMARY OUTCOMES:
To assess the efficacy of the transdermal system (TTS) as measured by the change from baseline in the frequency of total satisfying sexual activity captured by the Sexual Activity Log (SAL). | 2 years

SECONDARY OUTCOMES:
To assess the efficacy measured by the change from baseline in sexual desire using personal distress as measured by the Personal Distress Scale (PDS) score; the other 6 domains of the Profile of Female Sexual function, and the other 8 SAL endpoints. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Johna Lucas, MD, Study Director — Procter and Gamble
Locations (3):
- Research Facility, Chicago, Illinois, United States
- Research Facility, Randwick, Australia
- Research Facility, Québec, Quebec, Canada